CLINICAL TRIAL: NCT03917329
Title: An Evaluation of an ACT and PBS Group for Parents and Education Staff of Children and Young People With an Intellectual Disability
Brief Title: Evaluation of an ACT and PBS Group for Parents and Education Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 251260
Record Dates: First submitted 2018-11-06; First posted 2019-04-17 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Intellectual Disabilities With Other Behavioral Symptoms; Acceptance Processes; Psychological Distress; Burnout, Professional; Self Efficacy
Keywords: Parents; Education staff; Teachers; Intellectual Disability; Learning Disability; Positive Behaviour Support; Acceptance and Commitment Therapy; Group Therapy; Children; Psychological Distress
MeSH Terms: conditions — Behavior; Burnout, Professional; Intellectual Disability; Learning Disabilities

STUDY DESIGN:
Intervention Model Description: Participants will take part in a three session Acceptance and Commitment Therapy and Positive Behaviour Support group workshop and a focus group at a six week follow-up point. Pre-intervention, post-intervention and follow-up quantitative outcome questionnaire data will be gathered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT and PBS group workshop (Other): The intervention in this study is an Acceptance and Commitment Therapy (ACT) and Positive Behaviour Support (PBS) group workshop for parents and education staff of children with intellectual disabilities.
  Interventions: Other: ACT and PBS group workshop

INTERVENTIONS:
Other: ACT and PBS group workshop — Acceptance and Commitment Therapy and Positive Behaviour Support Group Workshop. Three sessions of approximately three hour duration. Groups will consist of 5-10 parents or 5-10 members of education staff. The group will include both didactic and experiential elements.

SUMMARY:
Parents and education staff who work with children with intellectual disabilities (ID) are known to be at a higher risk of experiencing psychological distress. This study evaluates whether a therapeutic group for parents and education staff who work with children with ID is effective in reducing psychological distress and if so, how it does this and who it works for. The group will include two components: an Acceptance and Commitment Therapy (ACT) section and a section about positive behaviour support (PBS). ACT is a psychological therapy, the aim of which is to help people to live their lives based on what matters to them, whilst learning new ways of managing difficult thoughts and feelings.

The PBS section aims to help participants to learn how to use positive strategies to reduce challenging behaviour. Both interventions have been shown to be effective on their own, but this study will examine if combining the two is helpful. Parents of children with ID and education staff who work closely with children with ID attending chosen schools or learning disability child and adolescent mental health services in NHS Lothian will be invited to participate in the study. The group will take place on three half days. Participants will complete questionnaires on the first and last day of the group and six weeks after it has finished. The questionnaires will be about psychological distress, confidence in caring for children with ID and seeing if the group changed how they cope with thoughts and feelings. Participants will also be invited to a focus group, which will think about if the intervention was helpful, and if so how it helped. If the group is effective, the investigators would hope to research the intervention in more depth with the aim of it being offered more widely in the future.

DETAILED DESCRIPTION:
Study Design

The study has a mixed methods design. The mixed methods approach allows the utilisation both quantitative and qualitative approaches to gain a greater level of detail than either one methodology would allow for individually, and for the results to support a firmer conclusion if the differing methodologies corroborate each other.

Protocol

The Learning Disability Child and Adolescent Mental Health Service (LD-CAMHS) service in NHS Lothian (National Health Service board located in Scotland) and schools for children with special educational needs in the City of Edinburgh Council area will be invited to participate in the study. Senior education staff (Headteachers or Deputy Headteachers) and LD-CAMHS clinicians will be asked to identify potential participants based on the study inclusion and exclusion criteria. They will then be asked to provide potential participants with the participant information sheet and discuss this with them, inviting potential participants to ask any questions that they may have. LD-CAMHS clinicians and education staff are suitable for this role as they are likely to be aware of children's diagnoses and whether the family have reported that their child presents with challenging behaviour, or aware of education staff's role and length of their remaining contract. Examples and a definition of challenging behaviour will be provided as a general guide to support the identification of participants. Interested potential participants will be given a minimum of 24 hours to consider whether they want to participate.

If interested in taking part, participants will be asked to complete and return a contact details form to their LD-CAMHS clinician or to senior education staff. The research team will contact the clinicians and senior education staff at agreed time intervals (e.g. once a week) to see if there are forms to be collected. In the contact details form, participants will be asked to indicate what time of day suits them best to be contacted. Participants will then receive a telephone call from the researcher to answer any questions they may have and to discuss their availability to attend the ACT and PBS group (e.g. would during or after school hours be preferable, are there certain days of the week that would suit them best, would location be a barrier).

Groups will aim to have 10 participants, with the expectation that some participants will choose to drop out of the study at this point, probably reducing the group size to approximately 6 to 8 participants. Participants will be allocated to attend a group based on their participant number, whether they are education staff or a parent, their location and availability. Participants will be sent a letter advising of the dates and location of their allocated group sessions and focus group. Should participants contact the researcher to advise that they cannot attend on these dates, they will be re-allocated to an alternative group if possible.

The ACT and PBS group will take place in a community setting such as an appropriate room in a school or in an NHS building. Participants will complete the study consent form with the study researchers on an individual basis before the first group session begins. This will provide a further opportunity for participants to ask any questions that they may have, and for the study researchers to ensure that participants are fully informed about the study and that they are making an informed decision to participate. Participants will then complete a battery of measures at the beginning of the first group session, at the end of the third group session and at the beginning of the focus group, which will take place six weeks after the last group session. Should a participant choose not to take part in the focus group, they will be sent a copy of the questionnaires by post and asked to return them by post via a returns envelope provided, or to their LD-CAMHS clinician or school.

The group workshop will run for three mornings, afternoons or evenings over three consecutive weeks (e.g. three Friday mornings). The sessions will last for approximately three to three and a half hours, with a break and refreshments in between. The group sessions will include taking part in exercises such as mindfulness, having group discussions, learning about new ways of managing difficult thoughts and feelings, and learning about new ways of supporting challenging behaviours in a positive way. Participants can decide not to take part in a component of the group should they prefer not to. Education staff and parents will attend separate groups. The group sessions will be facilitated by the study researchers, namely, a Trainee Clinical Psychologist and Clinical Psychologist who have both completed relevant ACT and PBS teaching and training and have experience in working with these psychological interventions.

The focus group will take place approximately six weeks later and will take approximately one hour in a similar setting as the therapy group. The group will be facilitated by a researcher who did not facilitate the participants' therapy group, to increase the likelihood that they will feel able to discuss the group freely. This researcher may be a LD-CAMHS clinician. The group will be audio-recorded with an NHS Lothian encrypted and password protected audio recorder, to allow for the group discussion to be transcribed and analysed. Participants who do not attend one or more of the group sessions will be welcome to attend the remaining sessions if they so wish but will be excluded from any relevant analyses. Participants may take part in the focus group if they have attended at least one group session.

Number of Participants

* The investigators will aim to recruit approximately 40 participants to the study (10 participants allocated to four groups).
* Number of sites involved: The investigators anticipate that there will be 8 (LD-CAMHS and up to 7 schools for children with special educational needs).
* Length of recruitment period: Estimated at approximately six to eight months.

Sample Size Calculation

Power calculations were performed utilising G-Power 3.1. The statistical analysis was set to be a with a within-between interaction, with two groups and three measurement points. The alpha level was set to 0.05 and power to 0.80, as per convention. The effect size previously reported for psychological distress in a similar study was medium to large. To be conservative, the power calculation for this study was performed with a medium effect size (f=0.25), which suggested a total sample size of 28 participants. Therefore, this study will aim to have four groups with ten participants each. This would mean recruiting 40 participants, with the expectation that 12 would be lost to attrition.

Proposed Analyses

The mean, standard deviation and range of the demographic variables and dependent variables will be reported. The percentage of missing data across the measures will also be reported.

Regarding quantitative data, the statistical analysis will be completed using SPSS software. Data will be explored to ensure that test assumptions are met. Each dependent variable will then be analysed with repeated measures analyses of variance (ANOVA) with a within-between interaction, with significant effects further evaluated appropriately.

Regarding qualitative data, the focus group interview transcripts will be analysed with thematic analysis.

Management of Missing Data

Should the level of missing data be minimal (<5%), the data will be assumed to be missing at random and a suitable method of imputation (most likely multiple imputation due to the small sample size) will be used to manage this appropriately. Should a higher level of missing data occur, the missing data will be analysed to examine whether it is missing at random or not. A suitable method of imputation will then be used.

Adverse Events

Should multiple participants present with high levels of persistent distress that appear to be related to participating in the group, this will be reviewed by the Chief investigator and researchers.

ELIGIBILITY:
Inclusion Criteria:

* Parent or Guardian of a Child aged 5-18 with a diagnosis of an Intellectual Disability/Learning Disability and experience of challenging behaviour.
* OR an employee working in a school for children with additional support needs, directly working with children with diagnosed Intellectual/Learning Disabilities.
* Must speak English fluently.
* Must be able to provide informed consent.

Exclusion Criteria:

* Temporary staff members (contract remaining of less than six months).
* Parents or Education Staff aged less than 18 years old.
* Parents or Education staff that have a diagnosis of an ID, such that they would not be able to understand the group materials or questionnaires and complete them independently.
* Individuals who are not able to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety and Stress Scale 21 item (DASS-21) | Pre-intervention (day 1, immediately before first group session), Post-intervention (at two weeks, day 15, at the end of the third group session) and at a six-week follow up (before the focus group).
  The DASS-21 is a 21 item outcome measure of psychological distress, and as such can measure change in psychological distress when multiple measurements are taken. The DASS-21 has three subscales of depression (range 0-21), anxiety (range 0-20) and stress (range 0-21), where higher scores are indicative of higher levels of psychological distress. The scores are multiplied by two to be comparable to the longer form of this measure, the DASS-42.

SECONDARY OUTCOMES:
Copenhagen Burnout Inventory (CBI) | Pre-intervention (day 1, immediately before first group session), Post-intervention (at two weeks, day 15, at the end of the third group session) and at a six-week follow up (before the focus group).
  The CBI is a 19 item outcome measure of burnout and as such measures changes in burnout. The CBI has three subscales of personal burnout (range 0-100), work related burnout (range 0-100), and client related burnout (range 0-100). In each subscale, scores 50-74 are indicative of moderate burnout, scores 75-99 are indicative of high levels of burnout, and a score of 100 is indicative of severe levels of burnout.
Comprehensive Assessment of Acceptance and Commitment Therapy Processes (ComPACT) | Pre-intervention (day 1, immediately before first group session), Post-intervention (at two weeks, day 15, at the end of the third group session) and at a six-week follow up (before the focus group).
  ComPACT is a 23 item outcome measure of ACT processes and as such measures changes in ACT processes over time. ComPACT has a range of possible scores between 0 and 138, where higher scores are indicative of higher levels of psychological flexibility. The measure has three subscales - openess to experience (range 0-60), behavioural awareness (range 0-30) and valued action (range 0 to 48).
Challenging Behaviour Self-Efficacy Scale (CBSES) | Pre-intervention (day 1, immediately before first group session), Post-intervention (at two weeks, day 15, at the end of the third group session) and at a six-week follow up (before the focus group).
  CBSES is a 5 item outcome measure of self-efficacy for managing challenging behaviour, and as such measures changes in this self-efficacy over time. The range of scores is 0 to 35, where higher scores are indicative of higher levels of self-efficacy for managing challenging behaviours in children with learning disabilities.

OTHER OUTCOMES:
Workshop Evaluation Measure (WEM) | Post-intervention (at two weeks, day 15, at the end of the third group session).
  The WEM is a 9 item outcome measure devised to evaluate the workshop. The WEM has five likert scale items and four free text open question items. The measure is likely to be examined item by item, rather than by items being summed. Higher scores in each item are indicative of higher levels of engagement or satisfaction with the workshop. Each likert scale item has a possible range of scores from 0 to 6.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Reid, MPsych, PhD, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - CAMHS-LD, NHS Lothian, Edinburgh, Midlothian
  - Edinburgh City Council, Edinburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative research in psychology, 3(2), 77-101.
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Cunningham, J. B., & McCrum-Gardner, E. (2007). Power, effect and sample size using GPower: Practical issues for researchers and members of research ethics committees. Evidence Based Midwifery, 5(4), 132-136.
- [Background] McConachie DA, McKenzie K, Morris PG, Walley RM. Acceptance and mindfulness-based stress management for support staff caring for individuals with intellectual disabilities. Res Dev Disabil. 2014 Jun;35(6):1216-27. doi: 10.1016/j.ridd.2014.03.005. Epub 2014 Mar 28. PMID 24685937

DOCUMENTS (3):
  • Informed Consent Form: Parent Consent Form (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT03917329/ICF_000.pdf
  • Informed Consent Form: Education Staff Consent Form (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT03917329/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT03917329/Prot_SAP_002.pdf